CLINICAL TRIAL: NCT04433780
Title: A Single Arm, Phase 3 Study, Exploring the Safety of Doravirine-based First-line Antiretroviral Therapy for Women of Reproductive Potential Living With HIV, a Pilot Switch Study Strategy in South Africa
Brief Title: DORA: A Doravirine-based First-line Antiretroviral Therapy for Women of Reproductive Potential Living With HIV
Acronym: DORA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Professor Francois Venter (Other)
Responsible Party: Sponsor-Investigator, Professor Francois Venter, Divisional Director of Ezintsha, University of Witwatersrand, South Africa
Organization: University of Witwatersrand, South Africa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EZMiM017
Record Dates: First submitted 2020-06-05; First posted 2020-06-16 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: HIV-1-infection
Keywords: Doravirine; Delstrigo; DOR/3TC/TDF; Women of reproductive potential
MeSH Terms: interventions — doravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Delstrigo (Experimental): Once-daily, fixed-dose combination of doravirine 100 mg, lamivudine 300 mg, and tenofovir disoproxil fumarate 300 mg (DOR/3TC/TDF).
  Interventions: Drug: Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate — DOR/3TC/TDF 100/300/300 mg once daily fixed-dose combination switched from either EFV/TDF/FTC or DTG/TDF/3TC
  Other Names: Delstrigo

SUMMARY:
This is a pilot study investigating the safety of Doravirine (DOR) in combination with Lamivudine (3TC) and Tenofovir Disoproxil Fumarate (TDF) administered over 48 weeks in women of reproductive potential living with HIV-1 switched from Efavirenz or Dolutegravir-based antiretroviral therapy on metabolic and neuropsychiatric outcomes.

DETAILED DESCRIPTION:
This is a pilot, open label, single-arm, single centre, phase 3, switch study exploring the safety of of Doravirine (DOR) in combination with Lamivudine (3TC) and Tenofovir Disoproxil Fumarate (TDF) administered over 48 weeks in women of reproductive potential living with HIV-1 switched from Efavirenz or Dolutegravir-based antiretroviral therapy. The metabolic and neuropsychiatric outcomes among women (and their infants) in a representative African female population of reproductive potential will be investigated.

Approximately 100 women aged between 18 and 49 years old will be administered a once-daily, fixed-dose combination of doravirine 100 mg, lamivudine 300 mg, and tenofovir disoproxil fumarate 300 mg (DOR/3TC/TDF). The study includes screening and baseline visits, 4 study visits from Week 4 to Week 36, and an end of study visit at Week 48.

ELIGIBILITY:
Inclusion Criteria:

* Females, aged 18-49 years and ≥ 40 kg
* On a first-line EFV or DTG-containing regimen for at least six months and not more than 3 years
* Plasma HIV-1 RNA < 50 copies/mL in last 60 days
* Calculated creatinine clearance (CrCl) > 50 mL/min (Cockcroft-Gault formula)
* Baseline weight measurement available at ART initiation.

Exclusion Criteria:

* Virological failure on any other regimen
* Women who are pregnant at the time of the screening or enrolment visits or have had a pregnancy gestation ≥ 28 weeks in the preceding 2 years
* Active tuberculosis and/or are on antituberculosis therapy at the time of the screening or enrolment visits
* Taking (and cannot discontinue) prohibited concomitant medications listed in protocol at least two weeks prior to the enrolment visit and for the duration of the study period (see potential drug interactions section for list).

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female HIV-positive participants of reproductive potential age
Enrollment: 133 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
The proportion of participants with neuropsychiatric adverse events (AEs) | 48 weeks
  The proportion of participants with neuropsychiatric adverse events (AEs) in 3 pre-specified categories (dizziness, sleep disorders/ disturbances, and altered sensorium) at Week 48
Changes in fasting lipids from baseline to Week 48 | 48 weeks
  Changes in fasting lipids from baseline to Week 48 assessed using lipid profile blood test
Changes in weight from baseline to Week 48 | 48 weeks
  Changes in weight from baseline to Week 48 assessed
Changes in body mass index from baseline to Week 48 | 48 weeks
  Changes in body mass index from baseline to Week 48 assessed
Changes in glucose from baseline to Week 48 | 48 weeks
  Changes in glucose from baseline to Week 48 assessed using blood test

SECONDARY OUTCOMES:
The proportion of participants with detectable plasma HIV-1 RNA levels (≥ 50 copies/mL) | At week 24, 48
  The proportion of participants with detectable plasma HIV-1 RNA levels (≥ 50 copies/mL) at weeks 24 and 48
The proportion of participants with neuropsychiatric adverse events (AEs) in 3 pre-specified categories | 24 weeks
  The proportion of participants with neuropsychiatric adverse events (AEs) in 3 pre-specified categories (dizziness, sleep disorders/ disturbances, and altered sensorium) at Week 24
Changes in glucose from baseline to week 24 | 24 weeks
  Changes in glucose from baseline to Week 24 using blood test
Changes in fasting lipids from baseline to week 24 | 24 weeks
  Changes in fasting lipids from baseline to Week 24 using lipid profile blood test
Changes in weight and from baseline to week 24 | 24 weeks
  Changes in weight from baseline to Week 24
Changes in body mass index from baseline to week 24 | 24 weeks
  Changes in body mass index from baseline to Week 24
The proportion of infants evaluated for HIV-positive tests using HIV DNA polymerase chain reaction test (PCR) | 48 weeks
  The proportion of infants evaluated for HIV-positive tests using HIV DNA polymerase chain reaction test (PCR)
Changes in quality of life from baseline | At weeks 24, 48
  Changes in quality of life from baseline to Weeks 24 and 48 measured using a traditional clinical, validated quality of life questionairre. Higher scores mean a better outcome
Median adherence by each adherence measure | At weeks 24, 48
  Median adherence by each adherence measure at Weeks 24 and 48 using a validated adherence questionairre
Emergence of antiretroviral resistance mutations in participants with virological failure | 48 weeks
  Evaluating the number of antiretroviral resistance mutations that emerge in participants with virological failure

CONTACTS AND LOCATIONS:
Overall Officials: Simiso Sokhela, Principal Investigator — Ezintsha, a subdivision of Wits Reproductive Health and HIV Institute (Wits RHI)
Locations (2):
- South Africa (2):
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng
  - Sunnyside Office Park, Johannesburg, Gauteng

IPD SHARING:
Plan to Share IPD: Yes
The data that will be shared is all of the individual participant data collected during the trial, after deidentification.The data that will be shared is all of the individual participant data collected during the trial, after identification. The data that will be shared is all of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication
Access Criteria: Anyone who wishes to access the data